CLINICAL TRIAL: NCT06945198
Title: Long-term Evaluation of Sports Activity in Patients Whose Ankle Was Treated by Anatomical Reconstruction or Arthroscopic Repair Following Chronic Lateral Instability
Acronym: ANKLE STAB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A02345-42; 2024-A02345-42 (Other: ANSM)
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Ankle Instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Broström's anatomical repair group (Active Comparator): Broström's anatomical repair is performed under arthroscopy. The principle of this method is to tighten and reattach the LTFA using very small anchors, when it is detached from the fibula but not too retracted and still of good quality. If necessary, this may also be accompanied by ligament reinforcement ('gould'), using a fragment of a fibrous structure in the ankle, the extensor retinaculum
  Interventions: Procedure: Broström anatomical repair
- Anatomical reconstruction group (Experimental): Anatomical ligamentoplasty or anatomical reconstruction is performed under arthroscopy. The principle of this method, which lasts around 40 minutes under spinal anaesthetic or general anaesthetic, is to reconstruct the LTFA and sometimes also the LCF, if it has been damaged, using a fragment of the tendon gracilis, located in the thigh, removed through an incision under the knee
  Interventions: Procedure: Anatomical reconstruction

INTERVENTIONS:
Procedure: Anatomical reconstruction — Anatomical ligamentoplasty or anatomical reconstruction is performed under arthroscopy. The principle of this method, which lasts around 40 minutes under spinal anaesthetic or general anaesthetic, is to reconstruct the LTFA and sometimes also the LCF, if it has been damaged, using a fragment of the tendon gracilis, located in the thigh, removed through an incision under the knee
  Arms: Anatomical reconstruction group
Procedure: Broström anatomical repair — Broström's anatomical repair is performed under arthroscopy. The principle of this method is to tighten and reattach the LTFA using very small anchors, when it is detached from the fibula but not too retracted and still of good quality. If necessary, this may also be accompanied by ligament reinforcement ('gould'), using a fragment of a fibrous structure in the ankle, the extensor retinaculum
  Arms: Broström's anatomical repair group

SUMMARY:
The goal of this clinical trial is to compare at 5 years the sporting activity of patients whose ankle had been treated by reconstruction or repair following chronic lateral instability. The main question it aims to answer is:

What is the long-term sporting activity status of patients whose ankle had been treated by reconstruction or repair following chronic lateral instability ?

Participants will visit the clinic once every year during 5 years for clinical checkup.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged ≥ 18 years
* Patient with chronic ankle instability defined by:
* A history of trauma including a severe ankle sprain.
* Clinical symptoms persisting for at least 3 months at the time of inclusion: pain, swelling, sensation of 'giving way', sensation of instability, recurrent sprains; Clinical tests (drawer test, varus provocation test) confirming grade III laxity; Imaging results (MRI) confirming clinically suspected ligament damage.
* Patient affiliated to or benefiting from a social security scheme
* French-speaking patient who has signed an informed consent form

Exclusion Criteria:

* Patient with deltoid ligament injury, severe fracture or open trauma
* Patient with insufficient ligament remnant and/or in too poor a condition to allow Broström-type repair.
* Patient with a symptomatic osteochondral lesion
* Patient with ankle hyperlaxity (Beighton score > 3)
* Patient with early ankle arthropathy (Takakura arthritis classification ≥ stage 3)
* Patient with neuromuscular disorders, systemic inflammatory disorders or tumours.
* Patient requiring surgery on both ankles
* Patients with a bony deformity of the ankle or foot on the affected side;
* Patients with professional athlete status
* Patient already included in another study
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Sporting activity | Year 5
  Patients' sporting activity will be assessed using the "Sport" subscale of the Quick FAAM (Foot and Ankle Ability Measure) questionnaire. Minimum value is 0 and maximum value is 32. 32 means a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France

IPD SHARING:
Plan to Share IPD: No